CLINICAL TRIAL: NCT02604381
Title: A Double Blind, Placebo Controlled Parallel Study on the Efficacy of Glucosamine Sulfate Potassium Chloride/Standardized Ginkgo Biloba Leaf Extract in Adults With Osteoarthritis of the Knee.
Brief Title: A Study on the Efficacy of Glucosamine Sulfate Potassium Chloride/Standardized Ginkgo Biloba Leaf Extract in Adults With Osteoarthritis of the Knee.
Acronym: 13GOHJ
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: KGK Science Inc. (Industry)
Collaborators: Joint Health Wellness Group, LLC. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 13GOHJ
Record Dates: First submitted 2015-11-10; First posted 2015-11-13 (Estimated); Last update posted 2017-08-11 (Actual); Status verified 2017-08

CONDITIONS: Osteoarthritis of the Knee
Keywords: Osteoarthritis; Knee; Glucosamine Sulfate; Ginkgo Biloba; WOMAC; Joint Health Wellness; Interleukin-1-beta
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Glucosamine Sulfate Potassium Chloride/Ginkgo Biloba Extract (Experimental): 2 capsules daily, immediately following a meal. 1 capsule in the morning, and 1 capsule in the evening, at approximately the same time each day.
  Interventions: Dietary Supplement: Glucosamine Sulfate Potassium Chloride/Standardized Ginkgo Biloba Extract
- Placebo (Placebo Comparator): 2 capsules daily, immediately following a meal. 1 capsule in the morning, and 1 capsule in the evening, at approximately the same time each day.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Glucosamine Sulfate Potassium Chloride/Standardized Ginkgo Biloba Extract
  Arms: Glucosamine Sulfate Potassium Chloride/Ginkgo Biloba Extract
Other: Placebo
  Arms: Placebo

SUMMARY:
The primary objective of the study is to assess the effectiveness of alpha-D Glucosamine Sulfate/Standardized Extract of Ginkgo Biloba Leaf versus a comparator product on osteoarthritis pain as assessed by the between group change in WOMAC™ Osteoarthritis Index Pain Subscale using Visual Analogue Scale (VAS) scores in subjects with osteoarthritis of the knee.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 45-70 years of age
* Body mass index (BMI) 18.0-39.9 kg/m2
* If female, subject is not of child bearing potential OR female subject of childbearing potential must agree to use a medically approved method of birth control and have a negative urine pregnancy test result.
* Primary or secondary, unilateral or bilateral osteoarthritis of the knee (American College of Rheumatology Clinical Criteria for Classification) characterized as knee pain with at least 3 of the following:
* Age > 50 years
* Stiffness < 30 minutes
* Crepitus
* Bony Tenderness
* Bony enlargement
* No palpable warmth
* Self reported difficulty performing at least one of the following activities because of knee pain:
* lifting and carrying groceries
* walking one-quarter of a mile
* getting in and out of a chair
* going up and down stairs
* mobility
* self-care activities
* Able to walk unassisted (may use walking stick, crutch, or knee brace)
* Availability for duration of the study period (2 week run-in +12 weeks)
* Subject agrees not to use over-the-counter medications or natural health products intended to treat OA pain during the run-in period and throughout the study (except the rescue medication provided).
* Subject using other therapies for OA, such as exercise, heat/cold therapy, joint protection and physiotherapy/occupational therapy agrees to continue these therapies as normal avoiding changes in frequency or intensity and to record therapies in the study diary
* Subject agrees not to start any new therapies for OA during the course of the study
* Agrees to maintain current exercise and dietary habits for the duration of the study
* Has given voluntary, written, informed consent to participate in the study

Exclusion Criteria:

* Women who are pregnant, breastfeeding, or planning to become pregnant during the course of the trial
* Physical examination findings show severe articular inflammation
* Subject has a diagnosis of rheumatoid arthritis, fibromyalgia, spinal disorders or other musculoskeletal disease
* Subject has been recommended for knee surgery
* WOMAC Pain Scale Score <4 for total pain (average of question #1 to question #5) at screening and baseline
* Subject has kidney or liver disease, blood disorders, active cancer and/or HIV infection
* Subjects with significant medical history or current metabolic disorders, thyroid disease, immune disorders and/or cardiovascular disease will be reviewed by the Qualified Investigator (QI). Subjects deemed by the QI to be at possible risk will not be permitted in this study.
* Subjects with a Type I or II diabetes
* Subjects with a history of seizures who are currently on medication to control seizures
* Subjects with hypertension will be reviewed by the Qualified Investigator (QI). If the subject is considered to be at risk they will not be permitted in this study
* Subjects with a history of reoccurring palpitations or dizziness
* Use of illicit drugs or history of drug or alcohol abuse with the past 2 years (currently having more than 2 standard alcoholic drinks per day)
* Planned surgery during the course of the trial
* Use of intra-articular, oral or parenteral corticosteroids, or other injectable prescription medication (e.g., Synvisc) within 2 months prior to randomization and during the trial
* Subjects taking prescription medication that affect blood coagulation (e.g. blood thinners, clotting factor replacements, acetylsalicylic acid)
* Subjects regularly taking over-the-counter medication (e.g. acetylsalicylic acid, ibuprofen) or natural health products (i.e. fish oils, vitamin E) that affect blood coagulation within 2 weeks of randomization
* Requires the use of prescription drugs to control pain (other than provided rescue medication)
* Use of oral or topical prescription or over the counter medications or natural health products for pain relief during the run-in period and during the trial (other than provided rescue medication, rescue medication should not be used within 72 hours prior to baseline and subsequent visits)
* Use of vitamins and minerals or natural health products/dietary supplements indicated for arthritis such as glucosamine and chondroitin sulfate within 2 weeks prior to the run-in period and during the trial
* Clinically significant abnormal laboratory results at screening (i.e. ≥ 2 times the ULN)
* Allergy or sensitivity to test product ingredients, including shellfish
* Allergy or sensitivity to acetaminophen, the rescue medication
* Individuals who are cognitively impaired and/or who are unable to give informed consent
* Any other condition which in the Investigator's opinion may adversely affect the subject's ability to complete the study or its measures or which may pose significant risk to the subject

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2015-11; Primary Completion 2017-06-19 (Actual); Study Completion 2017-06-19 (Actual)

PRIMARY OUTCOMES:
WOMAC™ Osteoarthritis Index Pain Subscale as a measure of Osteoarthritis pain | 12 weeks
  Assessed at screening and every visit.

SECONDARY OUTCOMES:
WOMAC™ Osteoarthritis Index Pain Subscale as a measure of Osteoarthritis pain | 12 weeks
  Measured at screening and every visit. Within group changes assessed
WOMAC™ Osteoarthritis Index Total Score as a measure of Osteoarthritis | 12 weeks
  Measured at screening and every visit
WOMAC™ Osteoarthritis Index Stiffness Score as a measure of Osteoarthritis stiffness | 12 weeks
  Measured at screening and every visit
WOMAC™ Osteoarthritis Index Physical Fuction Score as a measure of Osteoarthritis Physical Function | 12 weeks
  Measured at screening and every visit
Rand SF-36 questionnaire score as a measure of Quality of Life | 12 weeks
  Measured at every visit
Cartilage Oligomeric Matrix Protein (COMP) | 12 weeks
IL-1 Beta | 12 weeks
Amount of rescue medication used | 12 weeks

OTHER OUTCOMES:
Safety Blood Panel | Over 12 weeks
Blood Pressure | Over 12 weeks
Heart Rate | Over 12 weeks
BMI | Over 12 weeks
Incidence of Adverse Events | Over 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Tetyana Pelipyagina, MD, Principal Investigator — KGK Science Inc.
Locations (1):
- KGK Synergize Inc., London, Ontario, Canada